CLINICAL TRIAL: NCT04395027
Title: Iatrogenic Atrial Septal Defect Study
Brief Title: Iatrogenic Atrial Septal Defect Study (iASD)
Acronym: iASD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Administratively closed with IRB
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Tiberio Frisoli, Senior Staff, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13708
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Septal Defect, Atrial
Keywords: mitral valve intervention; iatrogenic septal defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Usual care (No Intervention): These patients will not have their iatrogenic septal defect closed.
- Device (Experimental): These patients will have their iatrogenic septal defect closed after the mitral intervention is completed.
  Interventions: Device: atrial septal defect closure

INTERVENTIONS:
Device: atrial septal defect closure — The iatrogenic septal defect will be closed in the usual manner
  Arms: Device

SUMMARY:
This is an open-label, randomized, controlled trial of iatrogenic atrial septal defect closure with the an atrial septal occluder versus usual care observation in patients post-mitral valve intervention requiring large bore transspetal access.

DETAILED DESCRIPTION:
This study is an open label, prospective, multicenter, non-randomized single-arm study to evaluate the safety and efficacy of the closing iatrogenic atrial septal defects in patients undergoing transcatheter mitral valve procedures using large sheaths.

A maximum of 5 Clinical Sites (referred to as "Sites" in the remainder of this document) in the U.S. Two hundred and ten patients will be enrolled in this study. The patients will randomized 1:2 device: control. The anticipated accrual rate is approximately 20 Subjects per month for a total accrual period of approximately 12-18 months.

Patients may be enrolled into the study provided all inclusion and no exclusion criteria are met as specified in Section 4. Subjects will be evaluated through hospital discharge and return for follow-up visits at 30 days, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 at the time of informed consent signature.
2. Capable of complying with Protocol requirements, including follow-up.
3. An Informed Consent Form signed by Subject or legal representative.
4. Patient has had successful reduction of mitral regurgitation to at most moderate regurgitation post-mitral-clip.

Exclusion Criteria:

1. Remaining mitral regurgitation of ≥ moderate-severe
2. Subject unable or unwilling to provide informed consent
3. Concomitant severe aortic valve disease
4. Dialysis
5. Pregnancy or intent to become pregnant
6. Life expectancy < 1 year
7. Active bleeding
8. Inability to follow up with 6-month timepoint due logistical concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
survival | 6 month
  Survival at 6 months

SECONDARY OUTCOMES:
survival | 1 year
  survival at 1 year
Freedom from heart failure hospitalization | 1 year
  Heart failure hospitalizations at 1 year
NYHA Functional Class | 1 year
  Symptom status at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Eng, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Marvin Eng, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided